CLINICAL TRIAL: NCT00374309
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Recombinant Ebola Adenoviral Vector Vaccine, VRC-EBOADV018-00-VP, in Healthy Adults
Brief Title: Experimental Vaccine for Prevention of Ebola Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 060237; 06-I-0237
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-05-05

CONDITIONS: Ebola Hemorrhagic Fever; Ebola Virus Disease; Ebola Virus Vaccines; Envelope Glycoprotein, Ebola Virus; Filovirus
Keywords: Hemorrhagic Fever; Healthy; Immunity; T -Cells; Filovirus; Healthy Volunteer; HV
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

INTERVENTIONS:
Drug: VRC-EBOADV018-00-VP

SUMMARY:
This study will determine if an experimental vaccine to prevent Ebola virus infection is safe and what side effects, if any, it causes. Ebola virus infection may range from mild to severe, and may cause breathing problems, severe bleeding, kidney problems and shock that can lead to death. The vaccine used in this study contains man-made genetic material similar to one part of the Ebola virus, which is designed to stimulate an immune response to the virus. The vaccine itself cannot cause Ebola virus infection because it does not contain any Ebola virus.

Participants are assigned to one of three groups as they enter into the study. Of the first 16 people in the study, 12 receive the lowest study dose of vaccine and 4 receive placebo (an inactive substance). If this dose is safe, then of the next 16 people who enter the study, 12 receive a higher dose of the vaccine, and the remaining 4 receive placebo. If this dose is safe, the final 12 people in the last group of 16 receive the highest study dose, and 4 receive placebo. The vaccine is given as a single injection in the arm on the day of enrollment.

Participants keep a diary for 5 days, recording their temperature, symptoms and any reaction at the injection site. They call a study nurse the day after vaccination to report how they feel, and they return to the clinic approximately six times for follow-up evaluations. These visits may include a check of vital signs, physical examination, blood and urine tests, or other medical tests if needed.

...

DETAILED DESCRIPTION:
Study Design:

This is a Phase I, randomized, placebo-controlled, double-blinded study to examine safety, tolerability and immune response of a recombinant Ebola adenovirus serotype 5 vector (Ebola-rAd5) vaccine in healthy adults. The hypothesis is that this vaccine will be safe and elicit immune responses to Ebola. The primary objective is to evaluate the safety and tolerability of the investigational vaccine VRC-EBOADV018-00-VP in healthy subjects. The secondary objectives include immunogenicity evaluations and adenovirus serotype 5 antibody titers (Ad5 Ab) at Weeks 0, 4, and 24. Exploratory evaluations include immunogenicity evaluations at Weeks 2, 12, and 48.

Product Description:

VRC-EBOADV018-00-VP is a recombinant product composed of two replication-deficient recombinant adenovirus serotype 5 (rAd5) vectors encoding for glycoprotein (GP), one from the Zaire strain and one from the Sudan-Gulu strain of Ebola. The final formulation buffer will be used as the diluent and as the placebo control (Crucell placebo). Injections will be administered intramuscularly (IM) by needle and syringe.

Subjects:

Healthy adult subjects ages 18 to 50 years old.

Study Plan:

Forty-eight subjects will receive a 1 mL intramuscular (IM) deltoid injection, via needle and syringe, of the study agent or placebo in a deltoid muscle as shown in the schema. Dose escalation will occur about three weeks after the last injection in the preceding dose group following an interim safety data review by a Data and Safety Monitoring Board (DSMB), provided that there are no significant toxicities. No more than one subject per day will be enrolled for the first 6 enrollments into each dosage group and the sixth subject enrolled must have 5 days (Group 1) or 14 days (Group 2 and Group 3) of follow-up before proceeding with further enrollments into that group.

Study Duration:

Subjects will be evaluated at 7 or more clinical visits during the 48 weeks after the study injection.

Study Endpoints:

The primary endpoint is safety and tolerability of the vaccine administered at doses of 2 x 10(9), 2 x 10(10) and 2 x 10(11) virus particles (VP) by IM injection. Secondary endpoints are immunogenicity as indicated by Ebola-specific antibody and cellular immune responses at Weeks 0, 4 and 24 and Ad5 antibody titer at Weeks 0, 4, and 24. Exploratory analyses of immunogenicity will also be conducted on stored samples collected at other timepoints including Weeks 2, 12 and 48.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must meet all of the following criteria:

1. 18 to 50 years old.
2. Available for clinical follow-up through Week 48.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to donate blood for sample storage to be used for future research.
7. In good general health without clinically significant medical history.
8. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than 40 within the 28 days prior to enrollment.

   Laboratory Criteria within 28 days prior to enrollment:
9. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men
10. White blood cells (WBC) equal to 3,300-12,000 cells/mm(3)
11. Differential either within institutional normal range or accompanied by site physician approval
12. Total lymphocyte count greater than or equal to 800 cells/mm(3)
13. Platelets equal to 125,000 - 400,000/mm(3)
14. Alanine aminotransferase (ALT) less than or equal to 1.25 upper limit of normal
15. Serum creatinine less than or equal to 1 x upper limits of normal (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males)
16. Normal urinalysis defined as negative glucose, negative or trace protein and no clinically significant blood in the urine.
17. Negative FDA-approved HIV blood test, at low risk of HIV exposure as assessed by behavioral risk interview, and amenable to HIV risk reduction counseling. [Note: Results of HIV ELISA will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study]
18. Negative hepatitis B surface antigen (HBsAg)
19. Negative anti-HCV and negative hepatitis C virus (HCV) PCR.
20. a PTT within institutional normal range and PT less than or equal to upper limit of institutional normal range.

    Female-Specific Criteria:
21. Negative beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential.
22. A female participant must meet one of the following criteria:

    * No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation, OR
    * Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 24 of the study, OR
    * Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 24 of the study by one of the following methods:
    * condoms, male or female, with or without a spermicide
    * diaphragm or cervical cap with spermicide
    * intrauterine device
    * contraceptive pills or patch, Norplant, Depo-Provera or any other FDA-approved contraceptive method
    * male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply.

Women:

1. Breast-feeding or planning to become pregnant during the first 24 weeks after enrollment.

   Subject has received any of the following substances:
2. Ebola vaccines or any recombinant adenoviral vector vaccine in a prior clinical trial.
3. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the past six months. [Note: that use of corticosteroid nasal spray for allergic rhinitis, topical corticosteroids for an acute uncomplicated dermatitis, or short-acting beta-agonists in controlled asthmatics are not excluded.]
4. Blood products within 120 days prior to HIV screening
5. Immunoglobulin within 60 days prior to HIV screening
6. Live attenuated vaccines within 30 days prior to initial study vaccine administration
7. Investigational research agents within 30 days prior to initial study vaccine administration
8. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration
9. Current anti-tuberculosis prophylaxis or therapy

   Subject has a history of any of the following clinically significant conditions:
10. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain
11. Idiopathic urticaria within the past 2 years
12. Autoimmune disease or immunodeficiency
13. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or parenteral corticosteroids.
14. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
15. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
16. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
17. Hypertension that is not well controlled by medication or blood pressure that is more than 145/95 at enrollment.
18. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bruising or bleeding difficulties with IM injections or blood draws, or use of anticoagulant medications.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
20. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt.
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject's ability to give informed consent.
24. A family history of pulmonary embolism associated with deep vein thrombosis without a known cause (such as hormonal contraceptive use or neoplasm) in a biologically related parent, sibling, child under the age of 60 years, or a family history of systemic lupus erythematosus in a biologically related parent, sibling, or child of any age.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48
Dates: Start 2006-09-05; Study Completion 2009-05-05

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AE's).

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays).

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Geisbert TW, Jahrling PB. Exotic emerging viral diseases: progress and challenges. Nat Med. 2004 Dec;10(12 Suppl):S110-21. doi: 10.1038/nm1142. PMID 15577929
- [Background] Meslin FX. Global aspects of emerging and potential zoonoses: a WHO perspective. Emerg Infect Dis. 1997 Apr-Jun;3(2):223-8. doi: 10.3201/eid0302.970220. PMID 9204308
- [Background] Okware SI, Omaswa FG, Zaramba S, Opio A, Lutwama JJ, Kamugisha J, Rwaguma EB, Kagwa P, Lamunu M. An outbreak of Ebola in Uganda. Trop Med Int Health. 2002 Dec;7(12):1068-75. doi: 10.1046/j.1365-3156.2002.00944.x. PMID 12460399